CLINICAL TRIAL: NCT03083353
Title: Isradipine Enhancement of Virtual Reality Cue Exposure for Smoking Cessation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-09-0150; 1R21DA049539-01 (NIH)
Record Dates: First submitted 2017-02-24; First posted 2017-03-20 (Actual); Results first posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Nicotine Dependence; Smoking, Cigarette; Smoking Cessation; Smoking Behaviors; Smoking Reduction; Craving
Keywords: nicotine; craving; virtual reality cue exposure; smoking relapse; immersive video environment; extinction enhancer
MeSH Terms: conditions — Tobacco Use Disorder; Cigarette Smoking; Smoking Cessation; Smoking; Smoking Reduction | interventions — Isradipine

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive isradipine (ISR) or placebo (PBO).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study capsules will be prepared containing: (a) 15 mg immediate release isradipine or (b) pill placebo consisting of Avicel microcrystalline cellulose powder (non-digestible pass-through). Isradipine and placebo capsules will be identical in appearance to maintain the double-blind. Individual doses will be dispensed to participants by blinded personnel 75 m prior to the first cue exposure session and patients will be asked to remain in the clinic until session time.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- isradipine (Experimental): Participants will receive 15mg of immediate release isradipine.
  Interventions: Drug: Isradipine; Behavioral: Cue Exposure
- placebo (Placebo Comparator): Participants will receive a placebo pill identical in appearance to isradipine.
  Interventions: Behavioral: Cue Exposure

INTERVENTIONS:
Drug: Isradipine — Isradipine will be administered 90 minutes prior to the initiation of cue exposure.
  Arms: isradipine
Behavioral: Cue Exposure — Participants will be exposed to visual smoking cues (i.e., immersive 360 degree video environments) delivered through consumer virtual reality headset and handle cigarette packs to activate and extinguish craving.

SUMMARY:
The proposed study represents a crucial and important stage in translating basic research to strategies for treating nicotine dependence. The investigation addresses an important public health issue by testing an intervention - informed by basic research - that may lead to a more effective and efficient treatment for smokers. The expected findings should provide initial effect size data for the addition of isradipine to an integrated psychosocial/behavioral and pharmacological smoking cessation intervention for smokers, and thus provide the necessary data for a large-scale follow-up trial.

DETAILED DESCRIPTION:
The current protocol will apply a pharmacologic augmentation strategy informed by basic research in animal models of addiction. Our goal is to evaluate the enhancing effect of isradipine, an FDA-approved calcium channel blocker, on the extinction of craving-a key mechanism of drug relapse after periods of abstinence. To activate craving robustly in human participants, we will use multimodal smoking cues including novel 360° video environments developed for this project and delivered through consumer virtual reality headsets. Adult smokers will take either isradipine or placebo and complete the cue exposure protocol in a double-blind randomized control trial. In order to test the hypothesis that isradipine will enhance retention of craving extinction, participants will repeat cue exposure in a medication-free state 24 h later. The study will be implemented in a primary care setting where adult smokers receive healthcare, and smoking behavior will be tracked throughout the trial with ecological momentary assessment.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years old;
2. Willing and able to provide informed consent, attend all study visits, and comply with the protocol;
3. Daily smoker for at least one year; and
4. Currently smoke an average of at least 5 cigarettes per day.

Exclusion Criteria:

1. Current diagnosis of a psychotic, eating, developmental or bipolar disorder, or significant suicide risk;
2. Current treatment for smoking cessation or use of other nicotine products, including e-cigarettes;
3. Exclusion criteria related to isradipine administration: (a) known allergy or sensitivity to isradipine, (b) hypertension, (c) congestive heart failure, (d) any type of liver disease, (e) current pregnancy, (f) women of childbearing potential who are not using medically accepted forms of contraception, (g) current use of Rifampin, which decreases the availability of calcium channel blockers, or of Tagamet, which can increase hypotensive effects and inhibit hepatic metabolism of isradipine, (h) any other significant medical condition that increases risk, as determined by the study physician;
4. Significant vision problems that would prevent engagement with the 360° video environment; and
5. Past six month substance use disorder, other than nicotine use disorder, assessed by structured interview.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cara C Young, Ph.D., Principal Investigator — University of Texas at Austin; Jasper AJ Smits, Ph.D., Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Protocol files are available on the The Open Science Framework page for this project
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Supporting information will be added as it becomes available.
Access Criteria: Available files are stored on the The Open Science Framework page for this project.
URL: https://osf.io/pk9yf/

REFERENCES:
- [Derived] Young CC, Papini S, Minami H, Morikawa H, Otto MW, Roache JD, Smits JAJ. Isradipine augmentation of virtual reality cue exposure therapy for tobacco craving: a triple-blind randomized controlled trial. Neuropsychopharmacology. 2024 Oct;49(11):1711-1718. doi: 10.1038/s41386-024-01872-9. Epub 2024 May 24. PMID 38789642

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from January 2020 to June 2023 with a pause from March 2020 to December 2020 resulting from pandemic-related restrictions on research
Pre-assignment Details: To be eligible for randomization, individuals had to abstain from smoking, starting 24 hours prior to the treatment visit. Prior to randomization at the treatment visit, individuals who reported smoking or had carbon monoxide level that exceeded 4 ppm were ineligible to participate that day but could reschedule.
Period: Overall Study
Arm/Group | Isradipine | Placebo
Started | 40 | 38
Completed | 36 | 34
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Isradipine | Placebo | Total
Number analyzed (Participants) | 40 | 38 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.10 (12.14) | 44.76 (10.12) | 42.88 (11.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 25 | 23 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 8 | 13
  Not Hispanic or Latino | 35 | 30 | 65
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 5 | 2 | 7
  White | 31 | 33 | 64
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 38 | 78
Education level [Count of Participants; unit: Participants]
  Graduate School | 4 | 6 | 10
  College Graduate | 14 | 14 | 28
  Partial College | 13 | 11 | 24
  High School Graduate | 7 | 7 | 14
  Partial High School | 2 | 0 | 2
Years of daily smoking [Mean (Standard Deviation); unit: years] | 20.53 (12.23) | 23.42 (11.32) | 21.94 (11.81)
Craving intensity to smoking cues [Mean (Standard Deviation); unit: units on a scale] — Cigarette craving intensity reported on a scale from 0-100 with 100 being the highest level of craving.
  units on a scale | 51.13 (3.73) | 60.39 (3.83) | 55.76 (3.78)

OUTCOME MEASURES:

1. Primary Outcome: Craving Intensity to Smoking Cues
Description: Primary outcome measures will be craving intensity to smoking cues based on a scale from 0 (No craving) to 100 (Intense craving).
Time Frame: The outcome is measured in a medication-free cue exposure session conducted 24 hours after medication administration
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Isradipine | Placebo
Number analyzed (Participants) | 40 | 38
units on a scale | 40.50 (3.54) | 50.44 (3.59)

ADVERSE EVENTS:
Time Frame: 48 hours
Description: Adverse events were collected during session 1 and session 2.
Arm/Group | Isradipine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/38
Other Adverse Events (participants affected / at risk) | 15/40 | 4/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Isradipine (N=40) | Placebo (N=38)
Headache (General disorders) | 11 (11) | 3 (3)
Heart racing (Cardiac disorders) | 2 (2) | 0 (0)
Upset stomach (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dizziness (General disorders) | 2 (2) | 0 (0)
Discomfort with virtual reality protocol (General disorders) | 0 (0) | 1 (1) — discontinued the study because of discomfort with the virtual reality-cue exposure therapy protocol

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-11-07): https://cdn.clinicaltrials.gov/large-docs/53/NCT03083353/Prot_SAP_ICF_000.pdf